CLINICAL TRIAL: NCT05168917
Title: EURECA (EUropeanRElapseCAlprotectin) Study - Calprotectin as Prediction Marker of Relapse in Patients With Quiescent Ulcerative Colitis
Brief Title: EURECA (EUropeanRElapseCAlprotectin) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DiaSorin Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: CLI-PR-1601
Record Dates: First submitted 2021-12-10; First posted 2021-12-23 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2022-01

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: Basal visit and follow up visits at 3,9,and 18 months in which stool specimens wil be collected.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Ulcerative colitis in clinical and endoscopic remission (Other): Patients with established diagnosis of ulcerative colitis (UC) in clinical and endoscopic remission defined as clinical score = 0 at enrollment with no endoscopy flare up may participate to follow up. Proctosigmoidoscopy to document endoscopic remission has to be foreseen. The patients' inclusion/exclusion criteria are based on the established diagnostic procedures for the UC, i.e. colonoscopy at the time of diagnosis, endoscopic evidence of remission and clinical significant findings.
  Interventions: Diagnostic Test: LIAISON Calprotectin

INTERVENTIONS:
Diagnostic Test: LIAISON Calprotectin — Immunoassay for fecal calprotectin measurement

SUMMARY:
This study will investigate the correlation of fecal calprotectin (FC) values to quiescent ulcerative colitis and to disease activity (relapse) as assessed by clinical data and endoscopy.

DETAILED DESCRIPTION:
The study is prospective with a longitudinal approach. About 200 patients will be followed every 3 to 12 months (at basal, 3, 6, 9 and 12 months alternating visits to telephone contacts) and subsequently for further 6 months in 3 different sites (competitive enrollment, 1site/country, Italy, France and Spain respectively). Fecal samples for immunoassays will be collected at follow up visits, stored frozen (-20°C) and sent to testing lab for their determination.

The following assessments are foreseen:

Clinical history and demography (screening), Proctosigmoidoscopy (basal), Hemochromo with WBC differential count, C-reactive protein (every 6 months from screening up to 12 months; relapse), Coagulation (screening) Specimen collection for fecal calprotectin determination (within 1-2 weeks from Informed Consent signature; for basal time point; every next 3 months from basal up to 12 months and at month 18; relapse), Coproculture for Salmonella, Shigella, E. Coli and Campylobacter (relapse), Pharmacological ongoing therapy, Mayo score (each time point; relapse)

ELIGIBILITY:
Inclusion Criteria:

* Adults,18 years and older, either genders
* Subject previously diagnosed with left-sided colitis or pancolitis based on endoscopy and, if available, confirmed by histological examination of biopsy taken during endoscopy
* Subject in clinical and endoscopic remission. Remission will be documented by proctosigmoidoscopy.
* Subject who may receive maintenance therapy as per current medical practice, e.g. mesalazine, corticosteroids, azathioprine, anti-TNF
* Availability of stool specimen for basal time point
* Subject willing and able to sign, the approved Informed Consent Form for this project in accordance with international and national regulations
* Subject able to understand and follow study procedures

Exclusion Criteria:

* Any subject that does not meet the inclusion criteria
* Subject with microscopic colitis
* Subject with Crohn's disease
* Subject with limited proctitis
* Subject with severe chronic disease affecting the possibility to comply with the study protocol (i.e. severe cardiovascular disease, renal or liver failure, neurologic disease, hematological disease and mental disorder)
* Subject who is regularly taking oral anticoagulants
* Subject who is currently pregnant or lactating
* Subject unable or unwilling to subscribe informed consent
* Subject unable or unwilling to perform required study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2017-06-02 (Actual); Primary Completion 2020-01-13 (Actual); Study Completion 2020-01-13 (Actual)

PRIMARY OUTCOMES:
Clinical Sensitivity and 95% Confidence Interval (exact method) | Through study completion, an average of 36 months
  Computed and compared to the clinical diagnosis
Clinical Specificity and 95% Confidence Interval (exact method) | Through study completion, an average of 36 months
  Computed and compared to the clinical diagnosis
Positive Predictive Value and 95% Confidence Interval (exact method) | Through study completion, an average of 36 months
  Computed and compared to the clinical diagnosis
Kaplan-Meier survival curve | Through study complete, an average of 36 months
  Percent variation from one time point to the following one will computed and compared to the disease evolution determined by the clinician for each subject. This curve will be used to determine the ability of the calprotectin value at the time of subject recruitment to predict the relapse.

SECONDARY OUTCOMES:
ROC Analysis and the relevant plots | Through study completion, an average of 36 months
  Analysis will determine if the assay was assigned with appropriate cut-off value

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Malesci, Professor, Study Director — Istituto Clinico Humanitas, Head of Gastroenterology Department
Locations (3):
- Centre Hospitalier Universitaire De Nancy (CHU de Nancy) Department Gastroenterology, Nancy, France
- Istituto Clinico Humanitas Centro IBD Diparimento di Gastroenterologia, Milan, Italy
- Centro Médico Teknon Gastroenterologia Adultos, Barcelona, Spain

REFERENCES:
- [Derived] Fiorino G, Danese S, Peyrin-Biroulet L, Sans M, Bonelli F, Calleri M, Zierold C, Pollastro R, Moretti F, Malesci A. LIAISON(R) Calprotectin for the prediction of relapse in quiescent ulcerative colitis: The EuReCa study. United European Gastroenterol J. 2022 Oct;10(8):836-843. doi: 10.1002/ueg2.12268. Epub 2022 Jul 4. PMID 35789124